CLINICAL TRIAL: NCT05573789
Title: Investigation of Mutations in DNA Damage Repair Genes and Other Actionable Molecular Aberrations as Biomarkers in Patients With Prostate Cancer
Brief Title: Tumor Molecular Profiling in Patients With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: NIPD Genetics (Unknown)
Responsible Party: Sponsor
Other Study IDs: TR19/9
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Metastatic Prostate Adenocarcinoma
Keywords: tumor molecular profiling; Mutations; homologous recombination repair; BRCA2; Prognostic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tumor blocks from patients with recurrent locally advanced, metastatic and/or high-grade operable prostate cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with prostate cancer: Patients with recurrent locally advanced, metastatic and/or high-grade operable prostate cancer and available formalin-fixed paraffin-embedded tumor tissue. Patients received treatment at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments of oncology. Tumor molecular profiling was performed.
  Interventions: Genetic: Tumor molecular profiling

INTERVENTIONS:
Genetic: Tumor molecular profiling — Tumor molecular profiling was assessed using the ForeSENTIA® Prostate panel developed by NIPD Genetic
  Other Names: Next-generation sequencing

SUMMARY:
The aim of the study was to evaluate the prevalence, the prognostic and predictive value of gene alterations in unselected patients with prostate cancer. Patients with histologically confirmed prostate cancer, treated at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments, were included. The presence of gene alterations was assessed using the ForeSENTIA® Prostate panel developed by NIPD Genetic.

DETAILED DESCRIPTION:
Data on tumor molecular profiling of European patients with prostate cancer is limited. The aim of the study was to evaluate the prevalence, the prognostic and predictive value of gene alterations in unselected patients with prostate cancer. Patients with histologically confirmed prostate cancer, treated at Hellenic Cooperative Oncology Group (HeCOG)-affiliated departments, were included. The presence of gene alterations was assessed using the ForeSENTIA® Prostate panel developed by NIPD Genetic. The primary endpoint was the prevalence of gene alterations in homologous recombination repair (HRR) genes. Secondary endpoint was overall survival.

ELIGIBILITY:
Inclusion Criteria:

Metastatic prostate cancer Recurrent prostate cancer Locally advanced prostate cancer High-risk operable prostate cancer Available FFPE tumor tissue

Exclusion Criteria:

Absence of tumor tissue available for analysis Lack of informed consent Lack of clinicopathological data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Study Population: Patients with recurrent locally advanced, metastatic and/or high-grade operable prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Time from diagnosis to the date of death, through the completion of the study

SECONDARY OUTCOMES:
Prevalence of somatic mutations in clinically relevant genes | 3 years
  Number of patients with somatic mutations

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Cooperative Oncology Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: No